CLINICAL TRIAL: NCT02199418
Title: Phase 2 Study of Weekly Paclitaxel in Combination With Cisplatin as Neoadjuvant Therapy for Locally Advanced Breast Cancer Patients
Brief Title: Addition of Cisplatin to Neoadjuvant Therapy for T Locally Advanced Breast Cancer
Acronym: SHPD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Lu, Director of Breast Surgery, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-BC-001
Record Dates: First submitted 2014-07-14; First posted 2014-07-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Tubular Breast Cancer; Mucinous Breast Cancer; Invasive Ductal Breast Cancer; Inflammatory Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel and Cisplatin (Experimental): Paclitaxel: 80 mg/m² i.v. given weekly on day 1 q day 8 for 16 weeks. Cisplatin: 25 mg/m² weekly on day 1 ,8,and 15 q day 28 for 4 cycles.
  Trastuzumab (only for human epidermal growth factor receptor-2(HER2)-positive patients): Loading dose: 4 mg/kg, Maintenance dose: 2 mg/kg, day 1 q day 8 for 16 weeks. Post-surgery: up to a total duration of 1 year
  Interventions: Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
Drug: Cisplatin

SUMMARY:
The investigators hypotheses that paclitaxel combined with cisplatin in a weekly-based regimen as neoadjuvant chemotherapy is effective and tolerable for locally advanced breast cancer.

DETAILED DESCRIPTION:
In this trial, all the patients will have weekly paclitaxel and cisplatin as neoadjuvant chemotherapy for 4 cycles. Patients with Her2 positive tumor will also receive the trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18years and ≤70 years
2. At least on measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST). Histologically confirmed invasive breast cancer, tumor size ≥2 cm, T2-4 N0-2M0
3. ER/PR/HER-2 and Ki-67 status detected on core biopsy. ER/PR positive is defined as >1% stained cells and HER2-positive is defined as immuno-histochemistry (IHC) 3+ or FISH ratio ≥ 2.0
4. No prior systemic or loco-regional treatment of breast cancer
5. ECOG 0-2
6. Adequate bone marrow function:WBC≥4.0×109/L, Absolute neutrophil count（ANC）≥1.5×109/L, Platelets（PLT）≥100×109/L, Hemoglobin（Hb）≥90g/L;aspartate aminotransferase(AST),Alanine aminotransferase (ALT)≤1.5 upper normal limit （UNL）, creatinine≤1.5 UNL, bilirubin≤1.5UNL
7. No obvious main organs dysfunction

Exclusion Criteria:

1. Unwilling or unable to use an acceptable method of contraception in 8 weeks (including 8 weeks) after final dose of test drug
2. Patient is pregnant or breast feeding
3. Inflammatory breast cancer and metastatic breast cancer
4. Any evidence of sense or motor nerve disorders
5. Patients with medical conditions taht indicate intolerant to neoadjuvant therapy, including uncontrolled cardiovascular disease, severe infection
6. Any concurrent malignancy other than breast cancer
7. Know severe hypersensitivity to any drugs in this study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pathological complete response of breast and lymph nodes | after 4 months preoperative treatment

SECONDARY OUTCOMES:
Tolerability and Safety | 4 months during neoadjuvant therapy
  Descriptive statistics for the treatment will be given on the number of patients whose treatment had to be reduced, delayed or permanently stopped
Clinical and imaging response | 4 months during treatment
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests. (sonography, mammography, or MRI) after treatment
regional recurrence free survival (RRFS) | 5 years
  RRFS is defined as the time period between registration and first event
local recurrence free survival (LRFS) | 5 years
  LRFS is defined as the time period between registration and first event
distant-disease- free survival (DDFS) | 5 years
  DFS is defined as the time period between registration and first event
overall survival (OS) | 5 years
  OS is defined as the time period between registration and first event

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wan C, Zhou L, Jin Y, Li F, Wang L, Yin W, Wang Y, Li H, Jiang L, Lu J. Strain ultrasonic elastography imaging features of locally advanced breast cancer: association with response to neoadjuvant chemotherapy and recurrence-free survival. BMC Med Imaging. 2023 Dec 21;23(1):216. doi: 10.1186/s12880-023-01168-2. PMID 38129778
- [Derived] Sun L, Yin W, Wu Z, Wang Y, Lu J. The Predictive Value of Pre-therapeutic Serum Gamma-glutamyl transferase in Efficacy and Adverse Reactions to Neoadjuvant Chemotherapy among Breast Cancer Patients. J Breast Cancer. 2020 Oct;23(5):509-520. doi: 10.4048/jbc.2020.23.e59. PMID 33154826
- [Derived] Wu Z, Zhang L, Xu S, Lin Y, Yin W, Lu J, Sha R, Sheng X, Zhou L, Lu J. Predictive and prognostic value of ZEB1 protein expression in breast cancer patients with neoadjuvant chemotherapy. Cancer Cell Int. 2019 Mar 29;19:78. doi: 10.1186/s12935-019-0793-2. eCollection 2019. PMID 30976202